CLINICAL TRIAL: NCT04924296
Title: A Multicentre, Randomized, Double-blind, Parallel, Placebo-controlled Phase II Study to Evaluate the Efficacy and Safety of fSHR-1314 in Adult Patients With Lupus Nephritis
Brief Title: A Phase II Study to Evaluate the Efficacy and Safety of SHR-1314 in Lupus Nephritis
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Suzhou Suncadia Biopharmaceuticals Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: SHR-1314-203
Record Dates: First submitted 2021-06-07; First posted 2021-06-11 (Actual); Last update posted 2021-06-11 (Actual); Status verified 2021-05

CONDITIONS: Lupus Nephritis
MeSH Terms: conditions — Lupus Nephritis

STUDY DESIGN:
Intervention Model Description: SHR-1314 subcutaneous administration, a multicentre, randomized, double-blind, parallel, placebo-controlled study
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Treatment group A (Experimental)
  Interventions: Drug: SHR-1314
- Treatment group B (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: SHR-1314 — SHR-1314 s.c. + Steroids
  Arms: Treatment group A
Drug: Placebo — Placebo s.c. + Steroids
  Arms: Treatment group B

SUMMARY:
To demonstrate the efficacy of SHR-1314 at Week 12 in subjects with proliferation lupus nephritis in terms of improvement of 24h UPCR, compared to placebo. The study will also assess the safety and tolerability of SHR-1314 in the patient population over the study period.

ELIGIBILITY:
Inclusion Criteria:

1. Chinese adult pts (18-65yr), Male or Female
2. BMI≥18 kg/m2 and ≤ 35kg/m2
3. Confirmed diagnosis of LN, renal biopsy report data is within 3-months prior to the date of ICF is first signed

   3.1 Biopsy-proven proliferative lupus nephritis Class III or Class IV, either with or without the presence of Class V, using the 2003 ISN/RPS criteria.

   3.2 24h UPCR ≥ 1 at screening.

   3.3 24h UPR ≥ 1.0 g/d，≤ 3.5 g/d.

   3.4 eGFR > 45ml/min/1.73m2.
4. SLEDAI-2K≥8.

Exclusion Criteria:

1. Significant medical Problems like myocarditis, pericarditis, severe manifestations of neuropsychiatric SLE (NPSLE)
2. Subjects who have previously treated by both CYC and MMF (or other forms of mycophenolate)
3. With a hHistory of using 60 mg/d prednisolone (or equivalent dose) for more than 3 months prior to Baseline
4. History of inflammatory bowel disease or have other ongoing active autoimmune diseases
5. Required management of acute or chronic infections within the past 8 weeks.
6. At screening, history or symptoms of malignancy of any organ system, treated or untreated, within the past 5 years, regardless of whether there is evidence of local recurrence or metastases.
7. History of congestive heart failure (New York Heart Association [NYHA] functional classification ≥III), cerebro-cardiovascular events, or serious bleeding events at screening and / or randomization that in the judgement of the Investigator prevents the subject from participating in the study.
8. History of depression and/or suicidal ideation or any suicidal behavior based on an assessment using the Columbina Suicide Severity Rating Scale (C-SSRS) at screening and baseline . The subjects will be exluded if any answer to question is "yes" in the questionnaire orare clinically judged by the investigator to be at risk for suicide
9. Receipt of any IL-17/IL-17R targeted therapy within the past year.
10. Those who have participated in any clinical study for any drug or medical device within 3 months before screening.
11. Tested positive for human immunodeficiency virus (HIV), hepatitis B, or hepatitis C.
12. All subjects will be tested for tuberculosis status using IGRA and X-ray test. Subjects with active or latent tuberculosis will be excluded
13. History of severe allergic reaction to contrast agents or biological medicines.Current drug or alcohol abuse or dependence.
14. History of severe allergic reaction to contrast agents or biological medicines.Current drug or alcohol abuse or dependence.
15. Pregnant or nursing..

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2021-06-28 (Estimated); Primary Completion 2021-12-25 (Estimated); Study Completion 2022-09-03 (Estimated)

PRIMARY OUTCOMES:
percentage change of 24 hours UPCR from baseline to Week 12. | at 12 weeks

SECONDARY OUTCOMES:
Percentage change of 24 hours UPCR from baseline to Week 24 | from baseline to Week 24
Percentage change of 24 hours UPCR from Week 12 to Week24 | from Week 12 to Week24
Percentage of participants achieving 24h UPCR <0.5 g/g at Week 12 and Week 24 | at Week 12 and Week 24
Percentage of participants achieving renal Complete Response at Week 12 and Week 24 | at Week 12 and Week 24
Percentage of pts achieving renal Partial Response at Week 12 and Week 24 | at Week 12 and Week 24
Change in PGA from baseline to Week 12 and Week 24 | from baseline to Week 12 and Week 24
Change in SLEDAI-2K from baseline to Week 12 and Week 24 | from baseline to Week 12 and Week 24